CLINICAL TRIAL: NCT05579561
Title: Is the Vegetarian Version of Therapeutic Carbohydrate Restriction as Effective as the Omnivore Version: In the Context of Remission of Type 2 Diabetes
Brief Title: Vegetarian Ketogenic Diet VS Omnivore Ketogenic Diet - Protocol of a Keto-vege Diet for Remission of Type 2 Diabetes
Acronym: DT2-OFF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: BloomedIn (Industry)
Collaborators: Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DT2-OFF
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus Type 2 in Obese; Hypertension; Diabetes Mellitus Type 2 With Hyperglycemia; Inflammation; Dysbiosis
Keywords: Diabetes Mellitus Type 2; Hyperglycemia; Inflammation; Dysbiosis; Obesity; ketogenic diet; carbs restriction
MeSH Terms: conditions — Hypertension; Inflammation; Dysbiosis; Diabetes Mellitus, Type 2; Hyperglycemia; Obesity | interventions — Diet; Equipment and Supplies

STUDY DESIGN:
Intervention Model Description: In a clinical study pilot project, compare vegetarian therapeutic carbohydrates restriction to the omnivore version, in the contexte of reverse type 2 diabetes symptoms
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vegetarian ketogenic diet (Experimental): Participants will be required to eat a diet that is very low in carbohydrates, moderate in vegetarian proteins, including fish and eggs, with added healthy fats
  Interventions: Other: Diet
- Omnivor ketogenic diet (Active Comparator): Participants will be required to eat a diet that is very low in carbohydrates, moderate in animal protein, with added healthy fats.
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Participants, in both groups, will be required to eat a diet that is very low in carbohydrates, moderate in protein, with added healthy fats. They will also have to breath in the device to estimate the level of different exhale gaz.
  Other Names: Device

SUMMARY:
Diabetes is one of the biggest public health challenges of the 21st century because of the costs associated with its management, which are estimated at more than three billion dollars per year in Quebec. This cost has been growing steadily for 20 years now. A person with controlled diabetes mobilizes three times more medical resources than a person without diabetes (Diabetes Quebec, 2009). This amount increases rapidly with the associated complications. Therapeutic carbohydrate restriction (in an omnivorous context) used specifically to control glycemia is being studied more and more, but has never been verified in a vegan context. Some studies show that a vegan diet could be an effective way to help type 2 diabetics (T2DM) to better manage their blood sugar. Thus, it is necessary to question whether these effects can be accentuated in the context of a low or very low carbohydrate diet. Numerous publications have highlighted the role of the gut microbiota in metabolic diseases, including T2DM. Analysis of the microbiome before and after dietary change combined with daily breath testing will tell us more about possible intolerances and the role of the microbiome in T2DM management. Given the novelty of these hypotheses and its absence in the literature, it is relevant to undertake a first pilot project with a smaller number of participants in order to obtain preliminary data that will allow us to define more precisely the research avenues for a subsequent study.

DETAILED DESCRIPTION:
In recent years, there has been an explosion in the prevalence of obesity and type 2 diabetes (T2DM) worldwide. Obesity, high blood pressure, excessive insulin secretion and other risk factors are precursors to serious or chronic health problems such as diabetes. Type 2 diabetes, which affects more than 8.1% of the Quebec population (2017-2018), has an average annual increase in prevalence of 3.3%, not to mention its devastating direct and indirect consequences on cardiometabolic health and its astronomical costs for the health system.This is now a global concern for which researchers, health experts, and physicians are working together to find practical solutions. In 2016, more than 3.8 million deaths were directly attributed to diabetes or high blood sugar. The number of indirect deaths related to diabetes, however, is difficult to estimate. Despite this, there are strong evidences that diabetes increases the risk of cardiovascular disease, stroke and kidney failure.

Many physicians around the world use low-carbohydrate or ketogenic diets to reverse T2DM. Dr. Evelyne Bourdua-Roy, of the Reversa Clinic, has been doing that since January 2017. Over 2000 patients have chosen the clinic to eat differently in order to learn to better manage their obesity, hypertension, type 2 diabetes and related comorbidities. As a result of the strategies proposed by the Reversa Clinic, many medications are regularly reduced or completely stopped as a result of the changes made in the patients' diet. This results in substantial savings for patients and the health care system. It also results in improved patient health (glycated hemoglobin [HbA1c], C-reactive protein [CRP], hypertension, etc.). New guidelines released by the American Diabetes Association, Diabetes Australia and Diabetes UK now recognize low and very low carbohydrate diets as secure and effective treatments to improve blood sugar levels and to help manage blood sugar variations and thus better manage this disease. With over 8% of the population affected by the disease, Diabetes Canada issued a statement to this effect in the spring of 2020.

The low-carbohydrate diet in an omnivorous context is being studied more and more, but has never been verified in a vegetarian context.

Several studies show that a vegan diet may be an effective way to help T2DM's better manage their blood glucose. Thus, one must question whether these effects can be accentuated in the context of a low or very low carbohydrate diet. Given the novelty of this hypothesis and its absence in the literature, it is relevant to undertake a first pilot project with a smaller number of participants in order to obtain preliminary data that will allow us to define more precisely the research avenues for a subsequent study.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* Under medication to treat type 2 diabetes
* Aged ≥ 18 years through 70 years

Exclusion Criteria:

* Type 1 diabetes
* Aged <18 years or >70 years
* Abnormal or low blood C-peptide by standard laboratory measurements.
* Have already initiated the change to ketogenic or vegan diet for more than 1 month.
* Pregnant or breastfeeding women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-05-11 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline HbA1c | Baseline and week 26
  Complete blood workup including the HbA1c , are done at the beginning and at the end of the 6 months to measure the improvement of glycated hemoglobin
Change from baseline CRP | Baseline and week 26
  Complete blood workup including the C reactive protein , are done at the beginning and at the end of the 6 months to measure the improvement of the CRP
Change from baseline of fasting insulin | Baseline and week 26
  Complete blood workup including the 14 hours fasting insulin , are done at the beginning and at the end of the 6 months to measure the improvement of insulinemia
Change from baseline of triglycerides | Baseline and week 26
  Complete blood workup including triglycerides , are done at the beginning and at the end of the 6 months to measure the improvement of the lipid profil

SECONDARY OUTCOMES:
Change in the digestive gaz exhale after meal | 90 min after each meal, during the first 2 months and the last 2 months
  Breath tests done after each meal to show the decrease in inflammation and indigestion via the concentration of certain gaz like N2
Change in the microbiome | Baseline and week 26
  Analysis of faeces (16-s) at the beginning and at the end, in order to see the changes on the population of bacteria colonies in the digestive tract

CONTACTS AND LOCATIONS:
Overall Officials: Andre Marette, Study Director — Institut universitaire de cardiologie et de pneumologie de Quebec
Locations (1):
- Elna Clinic, Saint-Mathieu, Quebec, Canada

REFERENCES:
- [Background] Diabetes Canada Position Statement on Low-Carbohydrate Diets for Adults With Diabetes: A Rapid Review. Can J Diabetes. 2020 Jun;44(4):295-299. doi: 10.1016/j.jcjd.2020.04.001. Epub 2020 Apr 24. No abstract available. PMID 32475469
- [Background] Goldenberg JZ, Day A, Brinkworth GD, Sato J, Yamada S, Jonsson T, Beardsley J, Johnson JA, Thabane L, Johnston BC. Efficacy and safety of low and very low carbohydrate diets for type 2 diabetes remission: systematic review and meta-analysis of published and unpublished randomized trial data. BMJ. 2021 Jan 13;372:m4743. doi: 10.1136/bmj.m4743. PMID 33441384
- [Background] Gurung M, Li Z, You H, Rodrigues R, Jump DB, Morgun A, Shulzhenko N. Role of gut microbiota in type 2 diabetes pathophysiology. EBioMedicine. 2020 Jan;51:102590. doi: 10.1016/j.ebiom.2019.11.051. Epub 2020 Jan 3. PMID 31901868
- [Background] Khazrai YM, Defeudis G, Pozzilli P. Effect of diet on type 2 diabetes mellitus: a review. Diabetes Metab Res Rev. 2014 Mar;30 Suppl 1:24-33. doi: 10.1002/dmrr.2515. PMID 24352832
- [Background] Rezaie A, Buresi M, Lembo A, Lin H, McCallum R, Rao S, Schmulson M, Valdovinos M, Zakko S, Pimentel M. Hydrogen and Methane-Based Breath Testing in Gastrointestinal Disorders: The North American Consensus. Am J Gastroenterol. 2017 May;112(5):775-784. doi: 10.1038/ajg.2017.46. Epub 2017 Mar 21. PMID 28323273
- [Result] Athinarayanan SJ, Adams RN, Hallberg SJ, McKenzie AL, Bhanpuri NH, Campbell WW, Volek JS, Phinney SD, McCarter JP. Long-Term Effects of a Novel Continuous Remote Care Intervention Including Nutritional Ketosis for the Management of Type 2 Diabetes: A 2-Year Non-randomized Clinical Trial. Front Endocrinol (Lausanne). 2019 Jun 5;10:348. doi: 10.3389/fendo.2019.00348. eCollection 2019. PMID 31231311
- [Result] Lin CL, Huang LC, Chang YT, Chen RY, Yang SH. Effectiveness of Health Coaching in Diabetes Control and Lifestyle Improvement: A Randomized-Controlled Trial. Nutrients. 2021 Oct 29;13(11):3878. doi: 10.3390/nu13113878. PMID 34836135
- [Result] Kahleova H, Matoulek M, Malinska H, Oliyarnik O, Kazdova L, Neskudla T, Skoch A, Hajek M, Hill M, Kahle M, Pelikanova T. Vegetarian diet improves insulin resistance and oxidative stress markers more than conventional diet in subjects with Type 2 diabetes. Diabet Med. 2011 May;28(5):549-59. doi: 10.1111/j.1464-5491.2010.03209.x. PMID 21480966
- [Result] Wang LL, Wang Q, Hong Y, Ojo O, Jiang Q, Hou YY, Huang YH, Wang XH. The Effect of Low-Carbohydrate Diet on Glycemic Control in Patients with Type 2 Diabetes Mellitus. Nutrients. 2018 May 23;10(6):661. doi: 10.3390/nu10060661. PMID 29882884